ncreasing African Immigrant's Breast Cancer Screening PI: Jamilia R. Sly, PhD

NCT04450264

Document Date: 6-13-2023

## THE MOUNT SINAI HEALTH SYSTEM ICAHN SCHOOL OF MEDICINE AT MOUNT SINAI RESEARCH INFORMATION SHEET

Study ID: STUDY-19-00114 Form Version Date: 13Apr2023

Study Title: Increasing African Immigrants' Breast Cancer Screening

Principal Investigator (Lead Researcher): Jamilia Sly, PhD

Physical Address: 17 East 102<sup>nd</sup> Street, New York, NY 10029

Mailing Address: 1425 Madison Icahn Bldg, Floor 3, Box# 1077, New York, NY 10029

Phone: (212) 824-7813

The purpose of this research study is to evaluate the feasibility, acceptability and impact of AWESOME (African Women Ending Stigma on Mammography Exams) – an educational program that has been designed to address the specific challenges that African-born women face in terms of completing breast cancer screening. You are being asked to take part in a research study because you: 1) are a woman, 2) were born in an African country, 3) can speak English and/or French, and 4) are at least 38 years old.

Participation in the research study is voluntary. You can agree to join or not. You can also say yes now, and change your mind later. Deciding not to be in the research study, now or later, will not affect your ability to receive medical care at Mount Sinai.

If you choose to take part, you will be asked to:

- 1) Attend one workshop, in person or online, that will provide information about breast cancer and breast cancer screening (e.g., how to have a mammogram, how often to go for a mammogram) to a group of women, followed by an interactive question and answer session. This will take about 40 minutes.
- 2) Fill out an anonymous, private survey, <u>right before</u> the workshop starts. Through this first survey, the study team will collect demographic information of participants (e.g., age, country of birth), basic information about previous experiences with breast cancer screening (e.g., year of last mammogram, if any was done before), and baseline understanding of breast cancer and breast cancer screening. This should take about 15 minutes.
- 3) Fill out an anonymous, private survey, <u>right after</u> the workshop is over. Through this second survey, the study team will assess any change in your understanding of breast cancer and breast cancer screening, as well as your opinion about the workshop (e.g., was it too long or too short?). This should take about 15 minutes.
- 4) Engage in a group discussion to make suggestions on how to improve the workshop. This should take about 20 minutes.

Your participation in this research study is expected to last 90 minutes. There are 64 people expected to take part in this research study.

Rev. 11.11.2022



Effective Date: 6/13/2023 End Date:2/15/2024

## THE MOUNT SINAI HEALTH SYSTEM ICAHN SCHOOL OF MEDICINE AT MOUNT SINAI RESEARCH INFORMATION SHEET

Study ID: STUDY-19-00114 Form Version Date: 13Apr2023

You can choose not to answer any question you do not wish to answer. You can also choose to stop taking the survey or participating in the other research activities at any time. You must be at least 38 years old to participate. If you are younger than 38 years old, please stop reading now and communicate to the study team that you cannot be part of the study.

The possible risks to you in taking part in this research are:

- Risk of feeling uncomfortable participating in a workshop revolving around breast cancer and breast cancer screening.
- Risk of feeling uncomfortable providing feedback and commentaries that express your opinion on how to improve the workshop to better serve the communities of African-born people living in the United States.
- Risk of loss of private information; this risk always exists, but there are procedures in place to minimize the risk.

The possible benefits to you for taking part in this research are:

Learning new information about breast cancer and breast cancer screening.

To protect your identity as a research subject, no identifiable information will be collected. In any publication about this research, your name or other private information will not be used.

There may be costs to you for taking part in this study, including transportation to and from the study visit, or childcare during the study visit. If you agree to take part in this study, you will be paid with a \$60 Target gift card for your time and effort. Payment will be provided at the end of participation in the study (i.e., after the educational program, all surveys, and the group discussion are complete).

If you have any questions about this research, please contact the Lead Researcher at (212) 824-7813. You can also call the Program for the Protection of Human Subjects Office at (212) 824-8200.

Rev. 11.11.2022



Effective Date: 6/13/2023 End Date:2/15/2024